CLINICAL TRIAL: NCT01007162
Title: Patient Satisfaction in the Critical Care Unit: A Qualitative Phenomenological Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Natalie Pattison, Royal Marsden NHS Foundation Trust
Other Study IDs: CCR3181
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Last update posted 2009-11-03 (Estimated); Status verified 2009-11

CONDITIONS: Patient Satisfaction in the Critical Care Unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
To explore issues patient experience and satisfaction with a sample of patients recently discharged from critical care.

DETAILED DESCRIPTION:
Patients' perceptions of their medical care are of increasing importance to educators, researchers, and clinicians. The emphasis on patient experience and satisfaction is consistent with the trend towards holding health care professionals accountable to their consumers. Our understanding and advancement of patients' experience and satisfaction with care forms a pivotal role in ensuring individuals engage with healthcare services, adhere to therapies, and maintain ongoing relationships with providers. Experiences are best explored using interview techniques such as phenomenological interviewing. In our study we propose to use a hermeneutic phenomenological approach. Phenomenology is a way of qualitatively exploring a person's experience and their personal meanings from those experiences. It is an approach that considers the structure of a person's subjective experience and explores areas that might be hidden. A phenomenological approach looks for patterns that are shared by particular instances or experiences. The evaluation of patient satisfaction and experience is based on valuing patients' subjective perception of an experience. In our study, a phenomenological approach will generate a comprehensive description of a phenomenon or lived experience (i.e. stay in the Critical Care Unit). We will interview a sample of patients to explore experiences and to gain their meanings of their stay in critical care. This will hopefully lead to thinking around ways of improving patient experiences, satisfaction and care.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients who were admitted to the Critical Care Unit at the Royal Marsden Hospital
* Patients who are not now at the End of Life or palliative.
* Adults (i.e. patients >18 years of age.
* Patients staying more than 24 hours.

Exclusion Criteria:

* Very short stay patients (<24 hours)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients who were admitted to the Critical Care Unit at the Royal Marsden Hospital
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Pattison, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom